CLINICAL TRIAL: NCT02896101
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Pimecrolimus Cream, 1% (Glenmark Pharmaceuticals Ltd) to the Marketed Product ELIDEL® (Pimecrolimus) Cream, 1% (Valeant Pharmaceuticals North America LLC) in the Treatment of Mild to Moderate Atopic Dermatitis (AD).
Brief Title: Study of Generic Pimecrolimus Cream, 1% in the Treatment of Mild to Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Pharmaceuticals Ltd. India (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLK-1601
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Atopic Dermatitis
Keywords: Mild to moderate
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pimecrolimus Cream, 1% (Experimental): Pimecrolimus Cream, 1 % (Glenmark Pharmaceuticals Ltd) topical application
  Interventions: Drug: Pimecrolimus Cream, 1%
- Elidel® (Active Comparator): Elidel® (Valeant Pharmaceuticals North America LLC) topical application
  Interventions: Drug: Elidel® (pimecrolimus) Cream
- Placebo (Placebo Comparator): Placebo of Pimecrolimus Cream, 1% (Glenmark Pharmaceuticals Ltd) topical application
  Interventions: Drug: Placebo of Pimecrolimus Cream, 1%

INTERVENTIONS:
Drug: Pimecrolimus Cream, 1%
  Arms: Pimecrolimus Cream, 1%
Drug: Elidel® (pimecrolimus) Cream
  Arms: Elidel®
Drug: Placebo of Pimecrolimus Cream, 1%
  Arms: Placebo

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multiple-Site Study to Evaluate the Therapeutic Equivalence of a Generic Pimecrolimus Cream, 1% (Glenmark Pharmaceuticals Ltd) to the Marketed Product ELIDEL® (pimecrolimus) Cream, 1% (Valeant Pharmaceuticals North America LLC) in the Treatment of Mild to Moderate Atopic Dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female subjects 12 years of age and older.
* Non-immunocompromised, with a clinical diagnosis of mild to moderate AD that has failed to respond adequately to other topical prescription treatments for atopic dermatitis, or for whom those treatments are not advisable.
* Confirmed diagnosis of AD for at least 3 months using the diagnostic features as described by Hanifin and Rajka.
* IGA score of 2 (mild) or 3 (moderate) and ≥ 5% BSA affected at baseline.

Exclusion Criteria:

* Active cutaneous bacterial, viral or fungal infection in any treatment area at baseline (e.g., clinically infected AD).
* Sunburn, extensive scarring or pigmented lesion(s) in any treatment area at baseline and history or presence of skin conditions that would interfere with evaluations.
* History or presence of Netherton's Syndrome, immunological deficiencies or diseases, organ transplant, HIV, diabetes, malignancy, malignant or pre-malignant skin conditions, serious active or recurrent infection, systemic immunosuppressive regimens, clinically significant severe renal insufficiency or severe hepatic disorders.
* Use within one month before baseline of 1) oral or intravenous corticosteroids, 2) UVA/UVB therapy, 3) psoralen plus ultraviolet A therapy (PUVA), 4) tanning booths, 5) non-prescription ultraviolet (UV) light sources, 6) immunomodulators or immunosuppressive therapies, 7) interferon, 8) cytotoxic drugs, 9) tacrolimus or 10) pimecrolimus.
* Use within 14 days before baseline of: 1) systemic antibiotics, 2) calcipotriene or other vitamin D preparations, or 3) retinoids.
* Use within 7 days before baseline of: 1) antihistamines, 2) topical antibiotics, 3) topical corticosteroids or 4) other topical drug products.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects in each treatment group with treatment success (i.e., a grade of clear or almost clear; a score of 0 or 1, within the treatment area) based on the IGA of Disease Severity at the end of treatment (Visit 3; Day 15 ± 3). | Day 15

SECONDARY OUTCOMES:
Change in severity score from baseline to Visit 3 of the four individual signs and symptoms of AD (i.e., erythema, induration/papulation, lichenification and pruritus). | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nikhil Sawant, Study Director — Glenmark Pharmaceuticals Ltd.
Locations (27):
- United States (27):
  - Investigational Site 4, Hot Springs, Arkansas
  - Investigational Site 22, Little Rock, Arkansas
  - Investigational Site 20, Anaheim, California
  - Investigational Site 13, Fremont, California
  - Investigational Site 26, Norco, California
  - Investigational Site 17, Doral, Florida
  - Investigational Site 9, Hialeah, Florida
  - Investigational Site 16, Miami, Florida
  - Investigational Site 18, Miami, Florida
  - Investigational Site 19, Miami, Florida
  - Investigational Site 25, Miami, Florida
  - Investigational Site 8, Miami, Florida
  - Investigational Site 12, North Miami Beach, Florida
  - Investigational Site 3, Ormond Beach, Florida
  - Investigational Site 7, South Miami, Florida
  - Investigational Site 10, Tampa, Florida
  - Investigational Site 24, Tampa, Florida
  - Investigational Site 14, West Palm Beach, Florida
  - Investigational Site 1, Arlington Heights, Illinois
  - Investigational Site 21, Lake Charles, Louisiana
  - Investigational Site 2, Silver Spring, Maryland
  - Investigational Site 11, Saint Joseph, Missouri
  - Investigational Site 27, East Windsor, New Jersey
  - Investigational Site 5, High Point, North Carolina
  - Investigational Site 23, Raleigh, North Carolina
  - Investigational Site 15, Cincinnati, Ohio
  - Investigational Site 6, Nashville, Tennessee